CLINICAL TRIAL: NCT03250351
Title: Effectiveness of Nerve Mobilization Techniques at Improving Upper Limb Morbidity Following Breast Cancer Surgery
Brief Title: Nerve Mobilization Techniques After Breast Cancer Surgery
Acronym: PT-ND-BC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Maria Torres Lacomba, Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12/2009
Record Dates: First submitted 2017-08-04; First posted 2017-08-15 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Two groups: Experimental group & Control group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: As masking techniques, the people responsible for randomization of intervention in each group, the evaluation of subjects and data collection, the analysis of data will be independent. Participants are also masked, since we think they are unable to distinguish between NDG and CG interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural mobilization group (Experimental): 3 to 5 days after surgery, the participants assigned to this group will receive 9 sessions of early physical therapy plus educational program (described in Torres Lacomba M) plus neurodynamic techniques consisting of neural tissue longitudinal glide using the Upper Limb Neurodynamic Test 1 (ULNT1), the neurodynamic test sequence for the median nerve, described by Butler and adapted by de la Rosa. With participants in the supine position, the shoulder was abducted and externally rotated, the scapula depressed, the forearm supinated, and the wrist and fingers extended. Mobilization was applied by depressing the scapula, flexing the elbow, and elevating the scapula, extending the elbow, within a pain-free range. The mobilization was applied for 2 minutes. Each session will be of 40 minutes approximately and will be held 3 sessions a week for 3 weeks.
  Interventions: Other: Neural mobilization group; Other: Control group
- Control group (Active Comparator): 3 to 5 days after surgery, the participants assigned to this group will receive 9 sessions of early physical therapy plus educational program (described in Torres Lacomba M). Each session will be of 40 minutes approximately and will be held 3 sessions a week for 3 weeks.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Neural mobilization group — See arm/group descriptions
  Arms: Neural mobilization group
Other: Control group — See arm/group descriptions

SUMMARY:
Objective: to determine nerve mobilization techniques effectiveness at improving shoulder disability in the early breast cancer postsurgical period, and whether the effect was maintained at 24-month follow up. Design: prospective randomized and single blind trial where participants will be randomly allocated into two groups by EPIDAT 3.1 software. Follow-up will be conducted through seven physical therapy assessments: one before surgery, the second one after surgery, the third one post-physical therapy intervention, the fourth one after three months, the fifth after six months and, the sixth one after twelve months, and the seven one after 24 months. Participants: one hundred and forty women, who are undergoing a unilateral breast cancer surgery with axillary lymph node dissection in the Breast Cancer Unit from "Príncipe de Asturias" Hospital. Intervention: Early physical therapy to control group and Early physical therapy plus nerve mobilization to intervention group during the three following weeks from surgery. Hypothesis: nerve mobilization helps brachial plexus sliding among its interface which improves shoulder disability the inner arm.

Key outcomes: pain, functional impairment, physical therapy, quality of life. Data analysis: quantitative variables through t-student test and qualitative variable though Chi test through by Statistical Package for the Social Sciences software.

DETAILED DESCRIPTION:
After giving their written informed consent, the participants will be summoned to perform the first assessment prior to surgery. Once participants will be discharged from hospital, approximately 3-5 days following the surgery, will be summoned to perform the second assessment. Those who will fulfil the selection criteria will be randomly allocated into two groups by an independent physical therapist. The experimental group will receive Early Physical Therapy plus neural mobilization and the control group will receive Early Physical Therapy. The same physical therapist will carry out all interventions for both groups. The physical therapist who will carry out the randomization process as well as the one who will perform the interventions will be the only two study members aware of group allocation. A third independent and blinded physical therapist will perform the assessments for all participants. Both physical therapists have more than fifteen years' experience in the treatment of breast cancer side effects. The ULNT1 will be perform to detect mechanosenstiviy-induced pain at presurgical and postsurgical assessments. The test sequence and the criteria will be followed to identify a positive test will reproduce from de study of de la Rosa.

In both groups, those women who will develop axillary web syndrome symptoms will receive an approach that aim at improving vascular tissue flexibility. If secondary lymphoedema will diagnose then complex decongestive physiotherapy will carry out.

ELIGIBILITY:
Inclusion Criteria:

* Women treated for unilateral breast cancer with surgery, including axillary lymph node dissection at the Department of Gynecology and Obstetrics of "Príncipe de Asturias" Hospital
* No contraindication to physical therapy
* Informed consent read, understood, and freely signed

Exclusion Criteria:

* Bilateral breast cancer
* Systemic disease (metastases)
* Infection
* Loco regional recurrence
* Chemotherapy as a neoadjuvant treatment

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Change of shoulder disability | 7 physical therapy assessments to evaluate change from surgery: At baseline, 7 days from baseline, 1 month, 3 months, 6 months, and 12 months from baseline
  It will be measured by SPADI spanish validated version.
Change of shoulder range of motion | 7 physical therapy assessments to evaluate change from surgery: At baseline, 7 days from baseline, 1 month, 3 months, 6 months, and 12 months from baseline 7th after 24 months after intervention.
  It will be measured by an inclinometer under the universal instructions and validated of the goniometry.
Change of strenght | 7 physical therapy assessments to evaluate change from surgery: At baseline, 7 days from baseline, 1 month, 3 months, 6 months, and 12 months from baseline
  It will be measured by a dynamometer under the universal instructions.
Change of pain intensity | 7 physical therapy assessments to evaluate change from surgery: At baseline, 7 days from baseline, 1 month, 3 months, 6 months, and 12 months from baseline
  To measure the intensity and get the information on the characteristics (type of feeling, duration, aggravating factors and mitigating, irritability, nocturnal behavior and activities with the UL ...) will be used a validated questionnaire shoulder Pain and Disability Index (SPADI). Contains a numerical scale to collect each answer. The possible answers are 0 to 10, with 0 being no distress and 10 present such difficulty that needs help. The result of the questionnaire is between 0 (no pain) and 80 (the most pain possible).
Change of health related quality of life | 7 physical therapy assessments to evaluate change from surgery: At baseline, 7 days from baseline, 1 month, 3 months, 6 months, and 12 months from baseline
  It will be measured by FACTB spanish validated version.

CONTACTS AND LOCATIONS:
Overall Officials: María Torres-Lacomba, PhD, Principal Investigator — University of Alcalá
Locations (1):
- María Torres-Lacomba, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torres Lacomba M, Yuste Sanchez MJ, Zapico Goni A, Prieto Merino D, Mayoral del Moral O, Cerezo Tellez E, Minayo Mogollon E. Effectiveness of early physiotherapy to prevent lymphoedema after surgery for breast cancer: randomised, single blinded, clinical trial. BMJ. 2010 Jan 12;340:b5396. doi: 10.1136/bmj.b5396. PMID 20068255
- [Background] de la Rosa-Diaz I, Torres-Lacomba M, Acosta-Ramirez P, Orive IG, Nee RJ, de la Villa-Polo P, Andres-Esteban EM, Sanchez-Sanchez B. Protective myoelectric activity at performing upper limb neurodynamic test 1 in breast cancer survivors. A cross-sectional observational study. Musculoskelet Sci Pract. 2018 Aug;36:68-80. doi: 10.1016/j.msksp.2018.05.003. Epub 2018 May 22. PMID 29860136
- [Background] Torres-Lacomba M, Prieto-Gomez V, Arranz-Martin B, Ferrandez JC, Yuste-Sanchez MJ, Navarro-Brazalez B, Romay-Barrero H. Manual Lymph Drainage With Progressive Arm Exercises for Axillary Web Syndrome After Breast Cancer Surgery: A Randomized Controlled Trial. Phys Ther. 2022 Mar 1;102(3):pzab314. doi: 10.1093/ptj/pzab314. PMID 35079831
- [Background] Torres-Lacomba M, Sanchez-Sanchez B, Prieto-Gomez V, Pacheco-da-Costa S, Yuste-Sanchez MJ, Navarro-Brazalez B, Gutierrez-Ortega C. Spanish cultural adaptation and validation of the shoulder pain and disability index, and the oxford shoulder score after breast cancer surgery. Health Qual Life Outcomes. 2015 May 23;13:63. doi: 10.1186/s12955-015-0256-y. PMID 26001890
- See also: Physiotherapy in women´s health research group — https://fisioterapia-saludmujer.web.uah.es/